CLINICAL TRIAL: NCT06993870
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Initial Efficacy of HBT-708 Monotherapy for Patients With Advanced Solid Tumors
Brief Title: Phase I Study of HBT-708 for Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBT-708-101
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Arm 1 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 1 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708
- Arm 2 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 2 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708
- Arm 3 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 3 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708
- Arm 4 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 4 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708
- Arm 5 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 5 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708
- Arm 6 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 6 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708
- Arm 7 (Experimental): Dose escalation will be conducted using an accelerated titration plus traditional 3+3 design. Dose Escalation includes 7 levels, Q3W IV. Dose extension will be carried out at the selected level. dose level 7 of HBT-708 Q3W i.v.
  Interventions: Drug: HBT-708

INTERVENTIONS:
Drug: HBT-708 — bispecific antibody
  Other Names: SSGJ-708

SUMMARY:
The purpose of this study will be to evaluate the safety, tolerability, and inital efficacy of HBT-708 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a study of HBT-708 monotherapy in advanced solid tumors. This study includes dose-escalation and dose-expansion cohort, with the accelerated titration combined 3+3 dose escalation method. The administration frequencies of HBT-708 is Q3W i.v. All cohorts will assess the efficacy and safety of the preset several dose levels of HBT-708 in advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18 years or older.
2. Histologically and/or cytologically documented advanced or measurable solid tumors.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancey > = 3 months.
5. Willingness to provide written informed consent for the study.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Subjects must have recovered (≤ Grade 1 or pretherapy baseline) from AEs due to previously administered therapies. (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to HBT-708 The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any treatment-emergent adverse event (TEAE) and dose-limiting toxicities | up to 24 months (every cycle visit, each cycle is 21 days)
  Adverse event were defined as the appearance of undesirable signs, symptoms, or medical conditions that occurred after informed consent.
Determine the maximum tolerated dose (MTD) and the maximum administration dose | up to 24 months (every cycle visit, each cycle is 21 days)
  Adverse events were defined as the appearance of undesirable signs, symptoms, or medical conditions that occurred after a participant provided informed consent.

SECONDARY OUTCOMES:
the plasma concentration of HBT-708 | Cycle1Day1, Cycle1Day2, Cycle1Day4, Cycle1Day8, Cycle1Day15; Cycle2 Day1; Cycle3 Day1, Cycle3Day2, Cycle3Day4, Cycle3Day8, Cycle3Day15; then Day 1 of every 2 cycles ( each cycle is 21 days)
  PK parameters will be calculated from the blood plasma concentrations of HBT-708 using standard noncompartmental PK methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No